CLINICAL TRIAL: NCT07109284
Title: A Single Arm, Multi-center Phase II Study of Neoadjuvant Therapy With Sacituzumab Tirumotecan (Sac-TMT) and KL-A167 for Early-stage, High-risk ER+/HER2- Breast Cancer (NeoSaciA)
Brief Title: SKB264 Combined With KL-A167 Neoadjuvant Therapy for Early-stage, High-risk ER+/HER2- Breast Cancer
Acronym: NeoSaciA
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Shuangyue Liu, Professor, West China Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SKB264-IIT-003
Record Dates: First submitted 2025-07-31; First posted 2025-08-07 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-07

CONDITIONS: ER+HER2- Breast Cancer
MeSH Terms: interventions — 18-O-demethylcervinomycin A2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Sacituzumab Tirumotecan + Tagitanlimab (Experimental): Participants receive Sacituzumab Tirumotecan every 2 weeks (q2w) in combination with Tagitanlimab every 2 weeks (q2w) for 18 weeks. In addition, participants receive an antihistamine, an H2 antagonist of investigator's choice, acetaminophen (or equivalent), and dexamethasone (or equivalent) per each drug's product label prior to sacituzumab tirumotecan infusions.
  Interventions: Biological: Sacituzumab tirumotecan; Biological: Tagitanlimab

INTERVENTIONS:
Biological: Sacituzumab tirumotecan — Sacituzumab tirumotecan 5 mg/kg, intravenously (iv), Q2W
  Other Names: SKB264; sac-TMT
Biological: Tagitanlimab — Tagitanlimab 900mg, intravenously (iv), Q2W
  Other Names: KL-A167

SUMMARY:
This study aimed to evaluate the efficacy and safety of SKB264 combined with KL-A167 as neoadjuvant therapy in early-stage high-risk ER+HER2- breast cancer patients.

DETAILED DESCRIPTION:
This is a single-arm, multi-center, phase II clinical trial to evaluate the efficacy and safety of SKB264 combined with KL-A167 as neoadjuvant treatment for early-stage high-risk ER+HER2- breast cancer. Eligible patients receive intravenous injections of 5mg/kg SKB264 and 900mg KL-167 every 2 weeks, with a total duration of 18 weeks for neoadjuvant therapy.

During neoadjuvant therapy, tumor assessments will be conducted every 6 weeks, followed by surgery after neoadjuvant therapy is completed. Following surgery, participants have the option to receive additional adjuvant therapy at the discretion of the treating physician. Participants will be followed at least every 6 months initially as per standard clinical practice.

The primary endpoint is to determine the pCR rate of SKB264 combined with KL-A167. Secondary endpoints include ORR, EFS, OS, and safety profile. Safety was evaluated by measuring the occurrence and severity of adverse effects by National Cancer Institute Common Terminology Criteria for Adverse Events, Version 5.0.

ELIGIBILITY:
Inclusion Criteria:

1. Females aged 18-70 years;
2. Pathologically confirmed invasive ductal breast cancer and untreated previously；
3. Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1;
4. Life expectancy ≥3 months;
5. Have at least 1 measurable disease defined by RECIST v1.1;
6. T1c-T2 (tumor size ≥2 cm), clinical node stage (cN)1-cN2, or T3-T4, cN0-cN2;
7. Has confirmed ER+/HER2-：ER≥1%、HER2 IHC 0、1+ or 2+/ISH-）;
8. Tumor Grade 3 of ductal histology, Or Tumor Grade 2 of ductal histology having an ER expression level percentage between 1-10%
9. Tissue or blood available for biomarker assessment;
10. Adequate organ function;
11. Patients with negative serum pregnancy test and those with fertility potential must agree to use effective contraception during the treatment period and for at least 3 months after the last dose of study drugs;
12. Patients must voluntarily participate in this study, sign an informed consent form, exhibit good compliance, and be willing to cooperate with follow-up procedures；

Exclusion Criteria:

1. Inflammatory BC；
2. Has multi-centric breast cancer (presence of more than 1 tumor in different quadrants of the breast).
3. Has bilateral invasive breast cancer.
4. Has metastatic (stage IV) breast cancer.
5. Has left ventricular ejection fraction (LVEF) of <50% or below the institution limit of normal, as assessed by echocardiogram (ECHO) or multigated acquisition (MUGA) scan performed at screening.
6. Has received prior treatment for breast cancer.
7. Has received prior therapy with an anti-programmed cell death protein 1 (anti-PD-1), anti-programmed cell death-ligand 1 (anti-PD-L1), or anti-PD-L2 agent or with an agent directed to another stimulatory or co-inhibitory T-cell receptor (e.g. cytotoxic T-lymphocyte-associated protein 4 [CTLA-4], OX 40, CD137).
8. Has received prior treatment for targeting TROP2 and/or topoisomerase I;
9. Patients who have had other malignancies within the past five years will be excluded from the study, with exceptions for those who have been successfully treated for cervical carcinoma in situ, skin basal cell carcinoma, or squamous cell carcinoma of the skin;
10. Has hypersensitivity to any of the components or excipients used in the study treatments.
11. History of allogeneic organ transplantation;
12. Patients with a history of non-infectious interstitial lung disease (ILD) or non-infectious pneumonia requiring steroid treatment, those currently diagnosed with ILD or non-infectious pneumonia, or those with suspected ILD or non-infectious pneumonia that cannot be ruled out by imaging at the time of screening, will be excluded. Additionally, patients suffering from clinically severe pulmonary damage due to pulmonary comorbidities will also be excluded. This includes, but is not limited to, any underlying pulmonary disease (such as pulmonary embolism within the past three months, severe asthma, advanced chronic obstructive pulmonary disease, restrictive lung disease, pleural effusion) or any autoimmune, connective tissue, or inflammatory conditions potentially affecting the lungs (such as rheumatoid arthritis, Sjögren's syndrome, sarcoidosis), as well as those who have undergone a pneumonectomy.
13. Patients with active autoimmune diseases requiring systemic treatment within the past two years will be excluded from the study. Systemic treatment does not include hormone replacement therapy, such as insulin therapy for Type 1 Diabetes, thyroid hormone replacement for hypothyroidism, or physiological doses of glucocorticoids for adrenal or pituitary insufficiency.
14. Patients with active infection requiring systemic therapy.
15. According to the investigator's judgment, there are concomitant diseases that seriously endanger the patient's safety or affect the patient's completion of the study, including but not limited to high blood pressure beyond the control of drugs, serious diabetes, active infection, etc.
16. Patients for whom participation in the study was deemed to be inappropriate by the investigator for any other reason were also excluded.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 55 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2028-01 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Pathological Complete Response (pCR) Rate (ypT0/Tis ypN0) | Up to approximately 6 months (Time of surgery)
  No microscopically detectable remnants of aggressive tumors in breast and axillary lymph nodes, ductal carcinoma in situ is allowed

SECONDARY OUTCOMES:
pCR Rate (ypT0/Tis) | Up to approximately 6 months (Time of surgery)
  No microscopically detectable remnants of aggressive tumors in breast, ductal carcinoma in situ is allowed.
Objective response rate (ORR) | Up to approximately 6 months (Time of surgery)
  The percentage of participants with CR or PR as the best response during the neoadjuvant treatment, based on RECIST v1.1.
Event-Free Survival (EFS) | Up to approximately 3 years
  The time from the first treatment to disease progression that: precludes surgery, results in a local or distant recurrence, results in a second primary malignancy, or death due to any cause whichever occurs first.
Overall Survival (OS) | Up to approximately 3 years
  The time from the date of first treatment to date of death due to any cause.
Adverse events (AEs) | Up to approximately 9 months
  Evaluated by NCI CTCAE (version 5.0) :
  1. The incidence, severity, and correlation with the investigational drug of adverse events (AE), treatment-related adverse events (TRAE), and serious adverse events (SAE);
  2. The number and proportion of subjects who reduced their dosage and stopped treatment due to the aforementioned adverse events;
  3. Study the changes in vital signs, physical examination results, and laboratory results before, during, and after treatment.

IPD SHARING:
Plan to Share IPD: No